CLINICAL TRIAL: NCT06091514
Title: Connected Cardiology to Control Cardiac Rythm
Acronym: C4R
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Action Research Group (Other); Hôpital Lariboisière Fernand Widal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP230642
Record Dates: First submitted 2023-10-16; First posted 2023-10-19 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation
Keywords: Connected Watch, Atrial Fibrilation (AF), Atrial Arythmia AA, Implantable Loop Recorder (ILR)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This clinical investigation is a comparative, one group, controlled study.
  Each patient represents its own control. Patients with an ILR already implanted for the detection of AF will receive a CS Medical Watch for a period corresponding to the period at risk of AF, up to 1 year maximum.
  For each patient, results obtained with the ILR device will be compared to results obtained with the CS Medical Watch device.
  During the conduct of the study, all medical decisions will be taken according to the ILR already implanted. No medical decision will be taken on CardiacSense System information collected during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort group (Other): Patients will be followed during a period ranging from 3 to 12 months depending on his period at risk of AF. This period will be defined at the inclusion visit. During this period, the patient will be followed as part of usual care, considering the medical informations given by the ILR device already implanted.
  During this period, the patient will have to wear the watch permanently outside charging time. Moreover, he will have to realize ECG measurement when the Medical Watch will indicate it. The patient could also trigger an ECG measurement if he feels the need.
  Interventions: Device: CS Medical Watch; Other: Specific questionnaire

INTERVENTIONS:
Device: CS Medical Watch — The Use of the CS Medical Watch during the participation period of the clinical investigation (between 3 and 12 months according to the period at risk of AF).
Other: Specific questionnaire — Specific questionnaire during the last study visit (takes place at M3 to M12 according to the period at risk of AF)

SUMMARY:
New-onset of atrial fibrillation (AF) and atrial arrythmia (AA) in general, is important as it exposes patients to stroke or other embolic complications not to mention the risk of heart failure. AF detection in high risk populations such as patients with a recent stroke or TIA or, symptomatic patients with multiple risk factors for AF, is performed with long-term electrocardiography monitoring using frequently implantable loop recorders (ILR). These recorders have their own limitations related to the invasive nature of the device implanted under the skin of the chest with limited acceptation by the patients. Smart watches appear as useful alternatives, but they need to be evaluated in an all-comer population of patients highly exposed to AF, different from the large population studies conducted in healthy young adults with a low incidence of AF. The unique features of CardiacSense Medical System suggest that we could have an accurate noninvasive detection of AF in a selected population very much exposed to the risk of atrial fibrillation, the most frequent atrial arrhythmia.

DETAILED DESCRIPTION:
Study design :

This clinical investigation is a comparative, non-randomised, one group, controlled study.

Each patient represents its own control. The study will envolve 400 participants

Hypothesis :

Our hypothesis is that CardiacSense Medical System is an effective, safe, and better accepted alternative for detecting atrial fibrillation (AF) in a high-risk population than implantable loop recorders (ILRs).

Population :

Any patient aged 18 years or more, with an ILR implanted for the detection of AF will be eligible. The time of implantation will not matter as long as the batteries work. Each patient will be proposed a CS Medical Watch for a period corresponding to the period at risk of AF.

Main objective :

To compare the performance of the CardiacSense Medical Watch by pulse plethysmography (PPG) only to the gold standard method of ILR monitoring, to detect AF that lasts 5 minutes or more, in a population of patients at high risk of paroxysmal AF.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or more
* Patient having signed free, informed, and written consent
* Patient presenting one of the following situations :
* Post-stroke or TIA patient with an already in place ILR
* Patient with symptoms evocative of AF (e.g. increased heart rate, chest pain) with an already in place ILR
* Post-PFO closure patient with an already in place ILR
* Patient in sinus rhythm treated for the prevention of paroxysmal AF with an already in place ILR
* Patient at high risk of AF (at the discretion of the investigator) with an already in place ILR
* Patient with a period of risk of AF ≥ 3 months.

Exclusion Criteria:

* Patient under legal protection
* Pregnant and/or breastfeeding women
* Patient with pacemakers, or ICD
* Patient with blood flow deficiency-related conditions
* Patient with tattoo or injured skin on the wrist
* Patient with tremors or otherwise unable to remain still for 15 minutes
* Patient without two hands and sufficient fingers to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The total number of episodes AF that lasts 5 min or more recorded on long-term monitoring | between 3 and 12 months according to the period at risk of AF
  The total number of episodes AF that lasts 5 min or more recorded on long-term monitoring using the CardiacSense Medical Watch by pulse plethysmography (PPG) only vs the gold standard method of ILR ECG recording, over the same period of monitoring by the two devices for each patient.

SECONDARY OUTCOMES:
The total number of AA episodes that lasts 5 min or more recorded on long-term monitoring | between 3 and 12 months according to the period at risk of AF
  The total number of AA episodes that lasts 5 min or more detected by PPG and confirmed by ECG measurement of the CardiacSense Medical Watch (vs. ILR ECG recording) over the same period of monitoring by the two devices for each patient.
The total number of episodes AF that lasts 5 min or more recorded on long-term monitoring | between 3 and 12 months according to the period at risk of AF
  Same primary endpoint for symptomatic patients vs. asymptomatic patients
The total duration of AF episodes that lasts 5 min or more | between 3 and 12 months according to the period at risk of AF
  Total duration of AF episodes that lasts 5 min or more / total duration of monitoring expressed in % for each device (PPG CS watch only vs. ILR ECG recording).
Incidence and severity of CS device vs ILR devices | between 3 and 12 months according to the period at risk of AF
  Related Adverse Events and incidents during the patient participation
Degree of invasiveness, comfort, and ease of use of both devices | between 3 and 12 months according to the period at risk of AF
  Description : measured using specific questionnaires for the study
Medico-economic evaluation according to the AP-HP hospital costs | between 3 and 12 months according to the period at risk of AF
  * The cost of each medical device (considering the replacement when needed over the study period for each patient)
  * The cost for extra-consultation/hospitalization for surgery, complication, or education.

IPD SHARING:
Plan to Share IPD: No